CLINICAL TRIAL: NCT01235351
Title: Escalating Clopidogrel by Involving a Genetic Strategy - Thrombolysis In Myocardial Infarction 56
Acronym: ELEVATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The TIMI Study Group (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIMI 56
Record Dates: First submitted 2010-11-02; First posted 2010-11-05 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: Myocardial infarction; Percutaneous coronary intervention; Clopidogrel; Genetics; Platelet Function
MeSH Terms: conditions — Myocardial Infarction | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel - for CYP2C19*2 carriers (Active Comparator): Clopidogrel for CYP2C19*2 gene carriers
  Interventions: Drug: Clopidogrel
- Clopidogrel - for CYP2C19*2 non-carriers (Active Comparator): Clopidogrel for CYP2C19*2 gene NON-carriers
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg daily, 150 mg daily, 225 mg daily, and 300 mg daily based on genotype
  Arms: Clopidogrel - for CYP2C19*2 carriers
Drug: Clopidogrel — Clopidogrel 75 mg daily, 150 mg daily
  Arms: Clopidogrel - for CYP2C19*2 non-carriers

SUMMARY:
To determine whether higher as compared with lower maintenance doses of clopidogrel can adequately improve the degree of platelet inhibition in carriers of a reduced-function CYP2C19 allele.

DETAILED DESCRIPTION:
Clopidogrel blocks the P2Y12 ADP receptor on platelets and has been shown to reduce cardiovascular events in acute coronary syndrome (ACS) patients.However, inter-patient variability in the pharmacodynamic response to clopidogrel is well recognized, and patients with lesser degrees of platelet inhibition in response to clopidogrel have been shown to be at increased risk of cardiovascular events.

One potential source of this variability is the metabolism of clopidogrel, which is a pro-drug requiring biotransformation to become an active antiplatelet compound. Cytochrome P-450 (CYP) enzymes play a role in the metabolism, and carriers of reduced-function genetic variants in CYP2C19 (~30% of the population) have lower active clopidogrel metabolite levels, diminished platelet inhibition, and higher rates of adverse cardiovascular events as compared with non-carriers in the setting of treatment with standard maintenance doses of clopidogrel.

Aim: To determine whether higher as compared with lower maintenance doses of clopidogrel can adequately improve the degree of platelet inhibition in carriers of a reduced-function CYP2C19 allele.

Hypotheses: The primary hypothesis is that subjects who carry a reduced-function CYP2C19 allele will have improvement in platelet inhibition with higher maintenance doses of clopidogrel.The secondary hypothesis is that higher maintenance doses of clopidogrel in carriers of a reduced-function CYP2C19 allele will result in similar platelet inhibition as compared to a standard maintenance dose of clopidogrel in non-carriers.

ELIGIBILITY:
Inclusion Criteria (major):

1. Between 18 and 75 years of age, inclusive.
2. Have an indication for the use of clopidogrel defined as either spontaneous MI [hospitalized with final diagnosis of MI, excluding periprocedural or definite secondary MI (e.g., due to anemia or hypertensive emergency)] or PCI within the past 6 months.
3. Clinically stable and at least 4 weeks following the MI or PCI.

Exclusion Criteria (major):

1. Conditions that alter platelet function.
2. Conditions that increase bleeding risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian T Ruff, MD, MPH, Principal Investigator — The TIMI Study Group
Locations (1):
- TIMI Study Group, Boston, Massachusetts, United States

REFERENCES:
- [Result] Mega JL, Hochholzer W, Frelinger AL 3rd, Kluk MJ, Angiolillo DJ, Kereiakes DJ, Isserman S, Rogers WJ, Ruff CT, Contant C, Pencina MJ, Scirica BM, Longtine JA, Michelson AD, Sabatine MS. Dosing clopidogrel based on CYP2C19 genotype and the effect on platelet reactivity in patients with stable cardiovascular disease. JAMA. 2011 Nov 23;306(20):2221-8. doi: 10.1001/jama.2011.1703. Epub 2011 Nov 16. PMID 22088980
- [Result] Hochholzer W, Ruff CT, Mesa RA, Mattimore JF, Cyr JF, Lei L, Frelinger AL 3rd, Michelson AD, Berg DD, Angiolillo DJ, O'Donoghue ML, Sabatine MS, Mega JL. Variability of individual platelet reactivity over time in patients treated with clopidogrel: insights from the ELEVATE-TIMI 56 trial. J Am Coll Cardiol. 2014 Jul 29;64(4):361-8. doi: 10.1016/j.jacc.2014.03.051. PMID 25060370
- [Result] Carreras ET, Hochholzer W, Frelinger AL 3rd, Nordio F, O'Donoghue ML, Wiviott SD, Angiolillo DJ, Michelson AD, Sabatine MS, Mega JL. Diabetes mellitus, CYP2C19 genotype, and response to escalating doses of clopidogrel. Insights from the ELEVATE-TIMI 56 Trial. Thromb Haemost. 2016 Jul 4;116(1):69-77. doi: 10.1160/TH15-12-0981. Epub 2016 Mar 24. PMID 27009617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 335 patients from 32 sites were enrolled from October 2010 until September 2011.
Pre-assignment Details: 335 patients enrolled, 2 patients not genotyped 333 patient allocated to initial treatment with 75 mg and 150 mg clopidogrel
Groups:
- CYP2C19*2 Non-Carrier: Period 1: clopidogrel 75 mg and 150 mg for 14 days each Period 2: crossover to sequences of clopidogrel (75 mg first, then 150 mg, and 150 mg first, then 75 mg) for 14 days each.
- CYP2C19*2 Carrier: Period 1: clopidogrel 75 mg and 150 mg for 14 days each Period 2: crossover to sequences of clopidogrel (225 mg first, then 300 mg, and 300 mg first, then 225 mg) for 14 days each.
Period: Initial Treatment With 75 mg and 150 mg
Arm/Group | CYP2C19*2 Non-Carrier | CYP2C19*2 Carrier
Started | 247 | 86
Completed | 237 (4 allocated to initial treatment included in primary analysis) | 82
Not Completed | 10 | 4
Not completed — No follow-up sample | 10 | 4
Period: Treatment With Different Dose Sequences
Arm/Group | CYP2C19*2 Non-Carrier | CYP2C19*2 Carrier
Started | 233 | 82
75 mg First and Then 150 mg | 116 | 0
150 mg First Then 75 mg | 117 | 0
225 mg First Then 300 mg | 0 | 41
300 mg First Then 225 mg | 0 | 41
Completed | 233 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYP2C19*2 Non-Carriers | CYP2C19*2 Carriers | Total
Number analyzed (Participants) | 247 | 86 | 333
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 60.8 (9.9) | 58.6 (9.7) | 60.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 23 | 84
  Male | 186 | 63 | 249

OUTCOME MEASURES:

1. Primary Outcome: Comparisons of Vasodilator-stimulated Phosphoprotein (VASP) Phosphorylation Platelet Reactivity Index (PRI)
Description: The outcome measurement was on-treatment PRI determined through flow cytometric assessment of phosphorylation status of VASP.
Time Frame: Approximately every 2 weeks for 8 weeks
Population: Non-carriers did not receive clopidogrel 225 mg or 300 mg
Measure: Mean (95% Confidence Interval); unit: % of PRI
Groups:
- CYP2C19*2 Carriers: Carrier of reduced function allele
- CYP2C19*2 Non-Carriers: Not a carrier of reduced function allele
Arm/Group | CYP2C19*2 Carriers | CYP2C19*2 Non-Carriers
Number analyzed (Participants) | 82 | 237
% of PRI
  Clopidogrel 75 mg: number analyzed (Participants) | 80 | 237
  Clopidogrel 75 mg | 71.0 [67.1 to 74.9] | 57.5 [55.1 to 59.9]
  Clopidogrel 150 mg: number analyzed (Participants) | 80 | 232
  Clopidogrel 150 mg | 62.4 [58.1 to 66.7] | 46.9 [44.3 to 49.1]
  Clopidogrel 225 mg: number analyzed (Participants) | 81 | 0
  Clopidogrel 225 mg | 54.0 [49.4 to 58.5] |
  Clopidogrel 300 mg: number analyzed (Participants) | 81 | 0
  Clopidogrel 300 mg | 50.1 [45.9 to 54.3] |

ADVERSE EVENTS:
Groups:
- CYP2C19*2 Carriers 75 mg: Patient with a carrier of genotype given 75 mg of the drug
- CYP2C19*2 Carriers 150 mg: Patient with a carrier of genotype given 150 mg of the drug
- CYP2C19*2 Carriers 225 mg: Patient with a carrier of genotype given 225 mg of the drug
- CYP2C19*2 Carriers 300mg: Patient with a carrier of genotype given 300 mg of the drug
- CYP2C19*2 Noncarriers 75 mg: Patients who are non-carriers of the genotype given 75 mg of the drug
- CYP2C19*2 Noncarriers 150 mg: Patients who are non-carriers of the genotype given 150 mg of the drug
Arm/Group | CYP2C19*2 Carriers 75 mg | CYP2C19*2 Carriers 150 mg | CYP2C19*2 Carriers 225 mg | CYP2C19*2 Carriers 300mg | CYP2C19*2 Noncarriers 75 mg | CYP2C19*2 Noncarriers 150 mg
Serious Adverse Events (participants affected / at risk) | 1/82 | 5/82 | 0/82 | 0/82 | 24/233 | 16/233
Other Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/82 | 0/82 | 0/233 | 0/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP2C19*2 Carriers 75 mg (N=82) | CYP2C19*2 Carriers 150 mg (N=82) | CYP2C19*2 Carriers 225 mg (N=82) | CYP2C19*2 Carriers 300mg (N=82) | CYP2C19*2 Noncarriers 75 mg (N=233) | CYP2C19*2 Noncarriers 150 mg (N=233)
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 1
Cardiac disorders (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 16 (16) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes